CLINICAL TRIAL: NCT02902536
Title: Tissue Repository for Studies of Myasthenia Gravis
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00078519
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — We will collect patient blood.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Myasthenia Positive Antibodies: Patients with Acetyl choline receptor (AChR) or muscle-specific kinase (MuSK) Positive Myasthenia
  Interventions: Other: No interventions
- Myasthenia Double Negative: Patients without AChR or MuSK antibodies
  Interventions: Other: No interventions
- Normal Controls: Patients without myasthenia
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions

SUMMARY:
This is a study during which the investigators collect plasma and cells from patients with myasthenia gravis for the purpose of finding new antibodies.

DETAILED DESCRIPTION:
This is a bio-specimen collection study. The investigators will collect plasma and peripheral lymphocytes. Plasma will be collected either when the patient undergoes plasma exchange, a decision independent of this study, or through a scheduled blood draw.

Patient plasma will be screened for novel antibodies which may cause myasthenia gravis. Subjects that are found to be positive for candidate antigens for myasthenia gravis will have a clinical evaluation which will consist of several disease rating scales will be performed (QMG score, MG-composite, Myasthenia Gravis Foundation of America (MGFA) clinical classification, MG-Quality of Life (QOL)15, MGFA Therapy Status).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Clinical Diagnosis of MG with supporting evidence either from antibody testing, repetitive nerve stimulations study (RNS) or Single Fiber Electromyography (EMG) (SFEMG).

Exclusion Criteria:

* Significant medical condition that would make participation in diagnostic and research part of evaluation impossible or risky. Acute or unstable medical condition.
* Inability to provide informed consent, either directly or via appointed power of attorney.
* Unwillingness to consent for collection of biological samples or their cryopreservation.
* Unable to provide evidence of previous antibody testing or neurophysiology confirming the diagnosis of Myasthenia Gravis.
* Any bleeding disorder that would prevent or present any danger during blood extraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Myasthenia Gravis and normal controls
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Identification of New Antibodies in Myasthenia Gravis assessed by enzyme-linked immunosorbent assay (ELISA) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No